CLINICAL TRIAL: NCT05966025
Title: Evaluation of the Potential Benefits of Itopride in the Management of Patients With Metabolic Associated Fatty Liver Disease
Brief Title: Potential Benefits of Itopride in the Management of Patients With Metabolic Associated Fatty Liver Disease (MAFLD)
Acronym: MAFLD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: October 6 University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Maha youssif, Maha Youssif Fekry, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-23006
Record Dates: First submitted 2023-07-14; First posted 2023-07-28 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Fatty Liver Disease; Fatty Liver
Keywords: Itopride in Mafld
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — itopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Experimental): • control group Weight reduction and life style modification(modification in diet like decrease lipids intak).pateints will recieve their conventional therapy
  Interventions: Drug: conventional therapy
- interventions: drug itopride (Experimental): • itopride group Weight reduction and life style modification and receive (itopride) 100 mg once dialy for 24 weeks plus their conventional therapy
  Interventions: Drug: Itopride; Drug: conventional therapy

INTERVENTIONS:
Drug: Itopride — itopride will be taken by pateints one time per day by dose 100 mg
  Arms: interventions: drug itopride
Drug: conventional therapy — will taken by patient in control group
  Other Names: Anti hypertensive druds, anti hyperlipidemic drugs

SUMMARY:
Objective of this study is to determine the clinical benefits of itopride in improvement of MAFLD

DETAILED DESCRIPTION:
the study will evaluate the possible benefits of itopride when added to pateints with metabolic associated fatty liver disease

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to hepatology clinic . -Patients are diagnosed by ultrasonography and laboratory tests for liver and lipids. - -
* Patients with comorbidites like hypertension,diabetes,dyslipidemia

Exclusion Criteria:

* Exclusion criteria included the presence of liver disease due to any of the following: viral hepatitis (HBV, HCV)
* acute systemic disease
* cystic fibrosis, coeliac disease
* suspicion of muscular dystrophy, alpha-1-antitrypsin deficiency
* metabolic inherited diseases
* autoimmune hepatitis, drug toxicity and drugs known to induce steatosis (e.g. valproate, amiodarone orprednisone).
* Patients were also excluded if body weight and carbohydrate metabolism were altered by the use of parenteral nutrition
* protein malnutrition
* previous gastrointestinal surgery
* structural abnormalitiesof the gastrointestinal tract or neurological impairment.
* the use of nonsteroidal anti-inflammatory drugs,antibiotics,sglt2,dpp4,statins,glp1
* probiotics or anti-secretory drugs capable of causing achlorhydria within 2 months preceding enrolmentwere also considered exclusion criteria.
* Patient with age below 18 or above 60

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-28 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
incidence of MAFLD | "1 Year "
  Highly sensitive CRP in mg\L by ELIZA, Fibro scan in MHzby fibroscan apparatus, ALT,AST in unit\liter by blood test

SECONDARY OUTCOMES:
Incidence of mafld | " 1 Year"
  Decrease LDL in mg\dl, Triglyceride and total cholesterolin mg\dl ,HOMA-IR in mg\dl, IL6,TNF alpha in mg\l by eliza

CONTACTS AND LOCATIONS:
Overall Officials: Hoda m rabea, A Professor, Principal Investigator — Beni-suaf university; Yasmine m madney, Lecturer, Principal Investigator — Beni-suaf university
Locations (1):
- Maha Youssif Fekry, Giza, Egypt